CLINICAL TRIAL: NCT02035540
Title: European Clinical Study for the Application of Regenerative Heart Valves - ESPOIR
Acronym: ESPOIR
Status: Completed | Type: Observational
Sponsor: corlife (Industry)
Collaborators: Hannover Medical School (Other); State University of Medicine and Pharmaceutics, Chisinau, Moldavia (Unknown); Leiden University Medical Center (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); University of Padova (Other); Hôpital Necker-Enfants Malades (Other); University of Zurich (Other); Universitaire Ziekenhuizen KU Leuven (Other); German Society for Tissue Transplantation (Other); European Homograft Bank (Other); Gottfried Wilhelm Leibniz Universität Hannover (Other)
Responsible Party: Sponsor
Other Study IDs: Surveillance Protocol 2013-11; FP7 2007-2013, No. 278453 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Heart Valve Disease
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Decellularized human valves: Pulmonary heart valve replacement
  Interventions: Other: Decellularized human valves

INTERVENTIONS:
Other: Decellularized human valves
  Other Names: ESPOIR PV

SUMMARY:
This is a prospective, non-randomized, single-arm, multicentre surveillance study to be conducted in Europe. The Surveillance is designed as a study, where

* ESPOIR pulmonary valve (PV) is prescribed in the usual manner in accordance with the terms of the approval.
* The assignment of the patient to a particular therapeutic strategy is not decided in advance by this Surveillance Protocol but falls within current practice and the prescription of ESPOIR PV is clearly separated from the decision to include the patient in the Surveillance.
* No additional diagnostic or monitoring procedures shall be applied to the patients
* and epidemiological methods shall be used for the analysis of collected data.

Evaluation of decellularized human heart valves for pulmonary heart valve replacement in comparison to current valve substitutes. Safety endpoints include cardiovascular adverse events, time to re-operation, re-intervention and explantation. Efficacy endpoints include freedom from valve dysfunction and hemodynamic performance.

ELIGIBILITY:
Inclusion Criteria:

* Indication for pulmonary valve replacement according to current medical guidelines in heart disease.
* Signed Informed consent of legal guardians or patients, assent of patients.

Exclusion Criteria:

* The patient has not provided Surveillance informed consent.
* The patient shall not suffer from

  * generalized connective tissue disorders (eg, Marfan syndrome), or
  * active rheumatic disorders, or
  * severe asymmetric calcification of the valve ring.
* The coronary arteries of the patient shall not be in abnormal position or heavily calcified.
* Patients shall not show hypersensitivity against Sodium Dodecyl Sulphate (SDS), Sodium Desoxycholate (SDC), human collagen (or other elastic fibers) or Benzonase®.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acquired and congenital heart disease requiring heart valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2014-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Amount of SARs (serious adverse reactions) | up to 24 months
  Cardiovascular Adverse Reactions; Serious Adverse Reactions, such as infections, immunological reactions, etc.
Freedom from valve dysfunction | up to 24 months
  Freedom from valve dysfunction leading to re-intervention or explantation at end of the study.

SECONDARY OUTCOMES:
Blood Parameters | up to 24 months
  Blood Parameters as additional safety data to support presence/absence of Adverse Reactions
Diameters of ESPOIR PV at end of the study | after 24 months
  Diameters of ESPOIR PV at end of the study in comparison to diameters at implantation
Time to reoperation | up to to 24 months
  Time to reoperation due to explantation
Time to death | up to 24 months
  Time to death
Evaluation of transvalvular gradients | up to 24 months
  valve competence assessed by noninvasive imaging tools such as echocardiography or cardiac magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Axel Haverich, Prof. Dr., Principal Investigator — Hannover Medical School; Samir Sarikouch, PD Dr., Study Director — Hannover Medical School
Locations (8):
- Universitair Ziekenhuis Leuven, UZL, Leuven, Belgium
- Université Paris Descartes, UPD, Paris, France
- Hannover Medical School, Hanover, Germany
- Università degli studi di Padova, Azienda Ospedaliera di Padova, UNIPD/AOP, Padua, Italy
- Universitatea de Stat de Medicina si Farmacie "Nicolae Testemitanu", SMPHU, Chisinau, Moldova
- Leids Universitair Medisch Centrum, LUMC, Leiden, Netherlands
- Universitaet Zuerich, UZH, Switzerland, Zurich, Switzerland
- Great Ormond Street Hospital for Children NHS Trust, GOSH, London, United Kingdom

REFERENCES:
- [Result] Boethig D, Horke A, Hazekamp M, Meyns B, Rega F, Van Puyvelde J, Hubler M, Schmiady M, Ciubotaru A, Stellin G, Padalino M, Tsang V, Jashari R, Bobylev D, Tudorache I, Cebotari S, Haverich A, Sarikouch S. A European study on decellularized homografts for pulmonary valve replacement: initial results from the prospective ESPOIR Trial and ESPOIR Registry datadagger. Eur J Cardiothorac Surg. 2019 Sep 1;56(3):503-509. doi: 10.1093/ejcts/ezz054. PMID 30879050
- [Result] Bobylev D, Horke A, Boethig D, Hazekamp M, Meyns B, Rega F, Dave H, Schmiady M, Ciubotaru A, Cheptanaru E, Vida V, Padalino M, Tsang V, Jashari R, Laufer G, Andreas M, Andreeva A, Tudorache I, Cebotari S, Haverich A, Sarikouch S. 5-Year results from the prospective European multi-centre study on decellularized homografts for pulmonary valve replacement ESPOIR Trial and ESPOIR Registry data. Eur J Cardiothorac Surg. 2022 Oct 4;62(5):ezac219. doi: 10.1093/ejcts/ezac219. PMID 35425983
- See also: ESPOIR Website — http://www.espoir-clinicaltrial.eu
- Available data/document: Study results — http://pubmed.ncbi.nlm.nih.gov/30879050/